CLINICAL TRIAL: NCT07061340
Title: The Effect of Therapeutic Touch on Agitation, Pain, and Cortisol Levels in Intensive Care Patients: A Randomized Controlled Study
Brief Title: The Effect of Therapeutic Touch on Agitation, Pain, and Cortisol Levels in Intensive Care Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/08-03
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Therapeutic Touch
Keywords: Therapeutic Touch; İntensive Care; Pain; Agitation; Cortisol; Nursing
MeSH Terms: conditions — Pain; Psychomotor Agitation | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Touch (Experimental): Therapeutic weaving will be done
  Interventions: Behavioral: Therapeutic Touch
- Control (No Intervention): Therapeutic weaving will not be done

INTERVENTIONS:
Behavioral: Therapeutic Touch — no Therapeutic Touch
  Other Names: Control
  Arms: Therapeutic Touch

SUMMARY:
Intensive care units (ICU) are special clinical areas where advanced monitoring and treatment of patients with life-threatening organ failure or those at risk of developing organ failure are carried out, with high technological equipment and a multidisciplinary approach is adopted. Agitation, pain, anxiety and hormonal imbalances are frequently observed due to hospitalization in ICU. In this stressful environment, patients often experience pain and agitation. Both situations trigger a physiological stress response in the patient and increase cortisol secretion. This increase in cortisol levels can suppress the immune system, delay wound healing and negatively affect the patient's general prognosis. Today, in addition to modern medicine, complementary/alternative therapies are increasingly used. One of these alternative therapies is therapeutic touch application. Therapeutic touch is based on the therapeutic effect of the act of touching. Therapeutic touch, alternatively known as healing touch, is a complementary/alternative treatment method applied by touching energy points on the body. Therefore, this study was planned to examine the effects of therapeutic touch applied to patients in intensive care on pain, agitation and cortisol levels. This study, planned as a randomized experimental study with a pre-test-post-test intervention control group, will consist of patients in the Intensive Care Unit of Fırat University Hospital. The sample will consist of 60 intensive care patients, 30 in the intervention group and 30 in the control group, who meet the research criteria on the specified dates and accept the research. The patients in the intervention and control groups will first be informed about the application before starting the application and their verbal and written consents will be obtained. Then, the intervention group will be given the Patient Identification Form, Richmond Agitation-Sedation Scale (RASS), Visual Analog Scale (VAS), cortisol levels from laboratory data will be recorded and therapeutic touch will be applied and after the application, the RASS and VAS scales will be filled again and the blood cortisol levels will be checked. This process will be done before and after each application and a total of 8 measurements will be taken. The application will take approximately 15-30 minutes every four days for the patients in the intervention group. During this period, no application will be made to the patients in the control group and RASS, VAS scales will be filled every four days and blood cortisol levels will be checked. Thus, a total of 8 measurements will be obtained. In the analysis of the data; frequency and percentage analyses, chi-square analysis, standard deviation, t-test in dependent groups, t-test analysis in independent groups will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and above.
* Patients who can communicate verbally.
* Patients who have been monitored in the intensive care unit for at least 4 days.
* Patients who are able to give informed consent.
* Patients who are hemodynamically stable.
* Richmond Agitation-Sedation Scale 1 and above.
* Visual Analog Scale 1 and above.

Exclusion Criteria:

1. Patients under deep sedation.
2. Patients on mechanical ventilation.
3. Patients with psychiatric problems.
4. Patients with skin diseases or open wounds, infections, burns that would prevent therapeutic touch.
5. Patients using sedative/analgesic drugs (excessive sedation or delirium).
6. Patients using corticosteroids or drugs that affect adrenal hormone levels (because these drugs can affect cortisol measurements).
7. Patients who have sudden life-threatening clinical changes during intensive care (e.g. sudden cardiac arrest, shock).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Richmond Agitation-Sedation Scale | After application,about 1 hour later
  The Richmond Agitation-Sedation Scale is a highly reliable and valid assessment tool developed to assess the agitation and sedation levels of intensive care patients. The scale is scored between -5 (deep sedation) and +4 (severe agitation) according to the patients' reactions to environmental stimuli. Individuals with a scale score of "0" are considered alert and calm, while negative scores indicate the depth of sedation and positive scores indicate the severity of agitation. It is widely preferred in clinical practice because it can be applied in a short time and can be used in an integrated manner with nursing care
Visual Analog Scale | After application,about 1 hour later
  The scale is frequently used in the assessment phase of pain intensity. Patients are asked to indicate the intensity of pain during activity or rest on a 10 cm long vertical or horizontal line. The line has a value of 0 at the beginning and 10 at the end. 10 means unbearable pain, and 0 means no pain at all. While the patient marks the pain they feel on this line, each point they mark is measured in cm.
Blood Cortisol Level | After application,about 1 hour later
  To be taken from patient records

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat university, Elâzığ, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No